CLINICAL TRIAL: NCT04261608
Title: A Retrospective Chart Review Study to Evaluate Safety of McGhan Single Lumen Gel-Filled Breast Implants in Patients in China
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MED-EPI-PLS-0637
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Breast Augmentation; Breast Reconstruction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a retrospective chart review and entails review of medical records of patients enrolled in about 5 hospitals/clinics in China, and who have undergone breast augmentation or reconstruction with McGhan breast implants between 24 December 2015 and 31 December 2019. The safety of McGhan breast implants (textured and smooth) will be evaluated based on occurrence of local complications including capsular contracture, malposition of implant, seroma/late seroma and anaplastic large cell lymphoma (ALCL).

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent breast augmentation or reconstruction with McGhan breast implants between 24 December 2015 and 31 December 2019

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Retrospective chart review study where data will be collected from all eligible patients who consecutively underwent breast implant surgery with McGhan single lumen gel-filled Breast implants from 24 December 2015 to 31 December 2019.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-07-04 (Actual); Study Completion 2020-07-04 (Actual)

PRIMARY OUTCOMES:
Number of participants who experienced adverse events | up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jie Luan, Professor, Principal Investigator — Chinese Academy of Medical Sciences
Locations (6):
- China (6):
  - Beijing Lidu Plastic Surgery Hospital, Beijing, Beijing Municipality
  - Plastic Surgery Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Guangzhou Sogood Medical Cosmetology Hospital, Guangzhou, Guangdong
  - The Second People's Hospital of Guangdong Province, Guangzhou, Guangdong
  - Changsha Yan Han Medical Plastic Hospital, Changsha, Hunan
  - Hunan Yamei Medical Cosmetology Hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: Yes
Allergan will share de-identified patient-level data and study-level data including protocols and clinical study reports for phase 2 - 4 trials completed after 2008 that are registered to ClinicalTrials.gov or EudraCT, have received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published. To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes. More information can be found on http://www.allerganclinicaltrials.com/.
Supporting Information: Study Protocol, CSR
Time Frame: After having received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published.
Access Criteria: To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes.
URL: http://www.allerganclinicaltrials.com/

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. — http://www.AllerganClinicalTrials.com
- See also: To be considered as a site for current and future Allergan Clinical Trials, please register using the Investigator Databank link. — http://www.investigatordatabank.org/